CLINICAL TRIAL: NCT04983784
Title: Buddhist Dalin Tzuchi General Hospital
Brief Title: The Effectiveness of Walking in Patients With Systemic Lupus Erythematosus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B10903020
Record Dates: First submitted 2021-07-09; First posted 2021-07-30 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Quality of Sleep; Quality of Life; Walking
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Sleep Initiation and Maintenance Disorders | interventions — Walking

STUDY DESIGN:
Intervention Model Description: The experiment group is composed of home walking, which contained walking guidance and telephone consultation, the control group without any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effectiveness of Walking on Sleep ,Depression and Quality of Life on intervention (Experimental): experimental group:
  1. intervention home-style walking exercises
  2. performed 12 weeks of 30 minutes walking exercise 2-3 times per week
  3. assess on at baseline and 12 weeks
  Interventions: Behavioral: walking
- No intervention group reaction (Experimental): control group:
  1. no intervention
  2. Routine care and follow-up
  3. assess on at baseline and 12 weeks
  Interventions: Other: Routine care

INTERVENTIONS:
Behavioral: walking — walking for 12 weeks at home
  Arms: The Effectiveness of Walking on Sleep ,Depression and Quality of Life on intervention
Other: Routine care — Routine care
  Arms: No intervention group reaction

SUMMARY:
Expected Results:

Finding from this evidence-based study ought to clarify the effectiveness of walking intervention for patients with SLE, and provide reference for future nursing strategies to improve disease adaptability.

DETAILED DESCRIPTION:
Background and purpose:

Walking exercise may be grateful in strengthening the cardiopulmonary function, regulating the joint flexbility, relieving the pain and the disturbance of sleep, all of which can further improve the quality of life among the patients with chronic diseases. Nevertheless, the information regarding the effect of walking exercise amongst systemic lupus erythematosus (SLE) subjects is still obscure. This study aimed to the influence of quality of life and sleep after the implementation of walking exercise among such groups.

uses the Psychometric evaluation of the Chinese version of the Pittsburgh Sleep QualityIndex、Systemic Lupus Erythematosus-Specific Quality of Life Questionnaire and Systemic Lupus Disease Activity of Lupus Erythematosus Disease Activity Score and Taiwanese Depression Questionnaire to evaluate the effectiveness of the intervention of walking exercise on Systemic lupus erythematosus.

Methods:

Through the quasi-experimental study design, the investigators intend to recruit the SLE patients from a hospital in Taiwan between 2021-2022. The main intervention is composed of home walking, which contained walking guidance and telephone consultation. After that, the investigators apply the structured questionnaires and existing data to collect performance indicators, covering the Chinese version of Pittsburgh Sleep QualityIndex, Systemic Lupus Erythematosus-Specific Quality of Life Questionnaire, Systemic Lupus Disease Activity of Lupus Erythematosus Disease Activity Score, and Taiwanese Depression Questionnaire. The effects of walking exercise is determined by The generalized estimation equations(GEE) .

ELIGIBILITY:
Inclusion Criteria:

* patients with fulfilled the American College of Rheumatology 1997 criteria for SLE

Exclusion Criteria:

* .patients with cardiovascular disease
* limited motion, such as bed-ridden, femur head necrosis
* were pregnant, or had a depressive disorder,

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
healthy quality of life Questionnaire | up to half a year
  The investigators will assess the Lupus Quality of Life(LupusQoL), from 0 (worst HRQOL) to 100 (best HRQOL)

SECONDARY OUTCOMES:
score system of depression | up to half a year
  The investigators will assess Taiwanese Depression Questionnaire (TDQ) The 18-item TDQ had a sensitivity of 0.89 and a specificity of 0.92 at a cutoff score of 19.
quality of sleep | up to half a year
  The investigators will assess Chinese version of Pittsburgh Sleep Quality Index (CPSQI) The CPSQI consists of 19 items that are used to generate seven component scores.
  A global CPSQI score > 5 indicates that patients suffer from sleep disturbance.

CONTACTS AND LOCATIONS:
Locations (1):
- Dalin Tzu Chi Hospital, Dalin, Taiwan